CLINICAL TRIAL: NCT05944042
Title: Hepatic Transplantation Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 002.HPB.2023.D
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-01

CONDITIONS: Identify More Accurate Predictive Models of Transplant Risk to Monitor and Evaluate New and Existing Patient Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intra-Operative Data:: Intra-Operative Data: Operative time, donor type, transfusions, intraoperative adverse events, mechanical ventilation, portal vein thrombosis, etc.
  Interventions: Other: Observational Transplant Analysis
- Post-Operative Data and Follow-Up:: Post-Operative Data and Follow-Up: Post-operative laboratories (MELD score, ctDNA, etc.), adverse events, discharge status, hospital length of stay, readmissions, recurrence of primary disease, graft survival, renal disease, post-transplant metabolic syndrome and major cardiovascular events, etc.
  Interventions: Other: Observational Transplant Analysis

INTERVENTIONS:
Other: Observational Transplant Analysis — Identify more accurate predictive models of transplant risk
  Other Names: Predictive models of transplant usage

SUMMARY:
The objective is to provide a mechanism to store information regarding the demographic characteristics; pre-, intra-, and post-transplant laboratories; treatment strategies; complications; and outcomes in patients undergoing hepatic transplantation.

DETAILED DESCRIPTION:
This study will be conducted at Methodist Dallas Medical Center and include data from hepatic transplant patients beginning in January 2019 and continuing until statistical significance is achieved. Patients will be identified based on ICD-10 procedure codes which are only available post-discharge in the EMR. Data will be collected once patient is discharged and no additional procedures are necessary. All cases meeting the inclusion criteria are expected to be included in this study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years Submitted to hepatic transplantation (Current Procedural Terminology® code 47135

Exclusion Criteria:

* Does not meet inclusion criteria specified in 3.1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age ≥18 years Submitted to hepatic transplantation (Current Procedural Terminology® code 47135 Patients will be identified based on ICD-10 procedure codes which are only available post-discharge in the EMR.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Need for prospective registry studies to determine patient factors to measure long-term survivial | 2 years
  As the demand for liver transplantation continues to grow, there is a need to identify more accurate predictive models of transplant risk. Therefore, prospective registry studies are needed to monitor and evaluate new and existing patient factors associated with long-term survival.
Methods of storing information on demographics of transplant patients | 2 yrs
  The objective is to provide a mechanism to store information regarding the demographic characteristics; pre-transplant, intra-transplant, and post-transplant laboratories; treatment strategies; complications; and outcomes in patients undergoing hepatic transplantation.

SECONDARY OUTCOMES:
Total Number and Description of Study Sites/Total Number of Subjects Projected | 2 yrs
  This study will be conducted at Methodist Dallas Medical Center and include data from hepatic transplant patients beginning in January 2019 and continuing until statistical significance is achieved. Patients will be identified based on International classification of Disease (ICD-10) procedure codes which are only available post-discharge in the EMR. Data will be collected once patient is discharged and no additional procedures are necessary. All cases meeting the inclusion criteria are expected to be included in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: Data can be access via the Methodist Health system Clinical Research Institute (Regulatory Department)

REFERENCES:
- [Background] Jadlowiec CC, Taner T. Liver transplantation: Current status and challenges. World J Gastroenterol. 2016 May 14;22(18):4438-45. doi: 10.3748/wjg.v22.i18.4438. PMID 27182155
- [Background] Zimmerman MA, Ghobrial RM, Tong MJ, Hiatt JR, Cameron AM, Hong J, Busuttil RW. Recurrence of hepatocellular carcinoma following liver transplantation: a review of preoperative and postoperative prognostic indicators. Arch Surg. 2008 Feb;143(2):182-8; discussion 188. doi: 10.1001/archsurg.2007.39. PMID 18283144